CLINICAL TRIAL: NCT06536647
Title: Contactless Assessment of Patient Vital Signs for Triage Using Remote Photoplethysmography in the Emergency Department - 1 Observational Study (CAPTURE-1 Study)
Brief Title: Contactless Assessment of Patient Vital Signs for Triage Using Remote Photoplethysmography in the Emergency Department
Acronym: CAPTURE-1
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: PanopticAI (Unknown)
Responsible Party: Sponsor
Other Study IDs: CAPTURE1
Record Dates: First submitted 2024-07-19; First posted 2024-08-05 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-07

CONDITIONS: Photoplethysmography; Vital Signs
Keywords: Photoplethysmography; Vital Signs; Emergency department; Triage
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Contactless measurement of patient vital signs using the VitalsTM system — Contactless measurement of the patient blood pressure, heart rate, respiratory rate, body temperature and SpO2 will be carried out using the VitalsTM platform based on facial video data.

SUMMARY:
Remote photoplethysmography (rPPG) is a camera-based method that enables contactless measurement of variation in light absorbance by haemoglobin as reflected by the changes in skin colour/pixel intensity unperceivable by human eyes. Beat-to-beat variation of light-absorbance can be used to estimate the change in the arterial blood volume underneath the skin and different vital signs including the blood pressure, heart rate, respiratory rate and oxygen saturation (SpO2) of the patient.

The investigators propose an observational prospective study to independently evaluate the accuracy of contactless vital sign measurements using a cell phone-based remote photoplethysmography (rPPG) technology. This study will recruit adult patients presenting to the Accident and Emergency Department (A&E) of Queen Mary Hospital (QMH) between 1 August 2024 and 30 October 2024. The study will be divided into 2 stages. In the initial run-in period, the investigators will collect facial video data from 200 patients to calibrate the VitalsTM system in the A&E environment. Then, the investigators will evaluate the accuracy of the VitalsTM in estimating vital signs of 1,000 ambulatory patients in the A&E setting.

A trained research nurse and research assistant will be deployed from 09:00 to 17:00 on weekdays to screen for eligible patients in the A&E waiting hall and to recruit patient participants throughout the study period. In this study, the investigators will only recruit triage category 3 (semi-urgent) to 5 (non-urgent) patients who are clinically stable and evaluate the performance of the VitalsTM in a designated room in A&E. Written informed consent will be obtained from all patient participants after an explanation of the details of the study, including the rationale, benefits and risks of participation.

After informed consent, contactless and manual measurement of patient blood pressure, heart rate, respiratory rate, body temperature and SpO2 will be carried out simultaneously in a designated room in A&E. A mounted light emitting diode (LED) will be used as the light source. Facial video of the patient participant will be captured using an iPhone, an iPad and a thermal camera placed at around 50 cm from the patient. A reference object for thermal and visual imaging will be placed at the background. Also, ambient temperature and light intensity will be measured.

The patient will be asked to sit down and remain still during video-recording. Manual measurement will be performed simultaneously by a trained research nurse or research assistant using standard hospital device or other medical-grade devices. A software program will be used to log vital sign measurements and recordings simultaneously so that data can be synchronised to reduce variations.

The primary outcome is the accuracy of the VitalsTM platform in estimating patient heart rate measured in intraclass correlation coefficient (ICC). The investigators will also measure of accuracy of the VitalsTM platform in estimating other vital signs, including blood pressure, respiratory rate, SpO2 and body temperature. The investigators will also evaluate patient satisfaction and comfort with the contactless and manual measurement techniques.

The accuracy of contactless measurement will be determined by calculating the ICC from the manual measurement readings as the ground truths. The investigators will also calculate the root mean square error (RMSE) and Pearson correlation between the contactless and manual measurement readings for individual vital signs. Altman Bland plot will be used to evaluate the bias and limits of agreement between two vital sign measurement methods.

ELIGIBILITY:
Inclusion Criteria:

* age >/= 18 years
* a valid written consent

Exclusion Criteria:

* age < 18 years
* refusal of consent/pre-existing mental illness rending consent impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a triage category 3 (semi-urgent) to 5 (non-urgent) rating who are clinically stable in the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The accuracy of patient heart rate estimation | 0 hour post-manual measurement
  The accuracy of the VitalsTM platform in estimating patient heart rate measured in intraclass correlation coefficient compared to manual heart rate measurement

SECONDARY OUTCOMES:
The accuracy of patient systolic blood pressure estimation | 0 hour post-manual measurement
  The accuracy of the VitalsTM platform in estimating patient non-invasive systolic blood pressure measured in intraclass correlation coefficient compared to manual systolic blood pressure measurement using a non-invasive cuff blood pressure device
The accuracy of patient diastolic blood pressure estimation | 0 hour post-manual measurement
  The accuracy of the VitalsTM platform in estimating patient non-invasive diastolic blood pressure measured in intraclass correlation coefficient compared to manual diastolic blood pressure measurement using a non-invasive cuff blood pressure device
The accuracy of patient respiratory rate estimation | 0 hour post-manual measurement
  The accuracy of the VitalsTM platform in estimating patient respiratory rate pressure measured in intraclass correlation coefficient compared to manual respiratory rate measurement
The accuracy of patient SpO2 estimation | 0 hour post-manual measurement
  The accuracy of the VitalsTM platform in estimating patient SpO2 measured in intraclass correlation coefficient compared to manual SpO2 measurement using a pulse oximetry
The accuracy of patient body temperature estimation | 0 hour post-manual measurement
  The accuracy of the VitalsTM platform in estimating patient body temperature measured in intraclass correlation coefficient compared to manual body temperature measurement using a thermometer
Patient satisfaction | Immediately after the measurements
  Patient satisfaction with the contactless and manual methods measured with a 10 cm visual analogue scale
Patient comfort | Immediately after the measurements
  Patient comfort with the contactless and manual methods measured with a 10 cm visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Rex Pui Kin Lam, MBBS, FHKCEM, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Accident and Emergency Department, Queen Mary Hospital, Hong Kong, None Selected
  - Accident and Emergency Department, Queen Mary Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Facial video data cannot be shared with other researchers according to the local patient privacy ordinance.
  Vital signs data from different measurement methods can be shared with other researchers upon reasonable request and after additional approval from the institutional review board.